CLINICAL TRIAL: NCT04032210
Title: The Influence of Preventive Regimens Containing Different Toothpastes on Caries Risk of High Risk Patients: A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Abdel Ghaffar Ahmed Ali, resident of conservative department of faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2230
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Prevention of Dental Caries
MeSH Terms: interventions — hydrated silica gel-based toothpaste; Crest Complete

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regimen using dual Zinc plus Arginine based toothpaste (Experimental)
  Interventions: Other: dual Zinc plus Arginine based toothpaste (Colgate total)
- Regimen using Zinc based toothpaste (Crest complete) (Experimental)
  Interventions: Other: Zinc based toothpaste (Crest complete)
- Fluoride based toothpaste (Signal) (Active Comparator)
  Interventions: Other: Fluoride based toothpaste (Signal)

INTERVENTIONS:
Other: dual Zinc plus Arginine based toothpaste (Colgate total) — Regimen using dual Zinc plus Arginine based toothpaste (Colgate total)
  Arms: Regimen using dual Zinc plus Arginine based toothpaste
Other: Zinc based toothpaste (Crest complete) — Regimen using Zinc based toothpaste (Crest complete)
  Arms: Regimen using Zinc based toothpaste (Crest complete)
Other: Fluoride based toothpaste (Signal) — Fluoride based toothpaste (Signal)
  Arms: Fluoride based toothpaste (Signal)

SUMMARY:
66 Participants will be divided into three groups according to the tested regimen (A), where (A1) represents participants will be exposed to regimen including dual zinc plus arginine based toothpaste (Colgate total), (A2) represents participants will be exposed to regimen including zinc based toothpaste (Crest complete) and (A3) represents control group where participants will be used fluoride based toothpaste (Signal). The study will be carried over a period of one year, assessment of cariogram will be done in two visits: first visit (baseline: T0) and second visit (after 3 months: T3) . In addition assessment of DMF scores will be done in four visits: first visit (baseline: T0), second visit (after 3 months: T3), third visit (after 6 months: T6) and final visit (after 12 months: T12) to obtain the required data

ELIGIBILITY:
Inclusion Criteria:

* • Normal adults will be recruited in this study, all the volunteers participated in this experiment will be healthy looking with free medical history.

  * Subjects of mean age 20-50 years.
  * Patients with high caries risk assessment according to Cariogram.
  * Non cariogenic diet patient
  * High plaque index
  * Not under antibiotic therapy either at the time of the study or up to the last month before the start of the study.

Exclusion Criteria:

* • Patients with a compromised medical history.

  * Cariogenic diet patient.
  * Participants with severe or active periodontal disease.
  * Participants with a history of allergy to any of the drugs or chemicals used in the study.
  * Patients on any antibiotics during the past month

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
caries risk assessment | Three months
  will be evaluated by cariogram

SECONDARY OUTCOMES:
DMF score | 12 months
  will be evaluated by ICDAS

CONTACTS AND LOCATIONS:
Locations (1):
- Esraa Abdel Ghaffar Ahmed, Giza, Other, Egypt

IPD SHARING:
Plan to Share IPD: Undecided